CLINICAL TRIAL: NCT06117865
Title: A Randomized Controlled Digital Intervention Study to Assess the Effect of Internet Delivered Interventions, the Low FODMAP-diet, Behavioral Therapy or Both, Compared to Patient Education, on Measures of Gastrointestinal Symptom Relief and Quality of Life in Patients With Irritable Bowel Syndrome
Brief Title: Digital Treatment of Irritable Bowel Syndrome (IBS)
Acronym: DIGIBS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-630038
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-05

CONDITIONS: IBS - Irritable Bowel Syndrome
Keywords: digital treatment
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Patient education (Sham Comparator)
  Interventions: Behavioral: Module 1; Behavioral: Module 2; Behavioral: Module 3
- Behavioral therapy (Active Comparator)
  Interventions: Behavioral: Module 1; Behavioral: Module 2; Behavioral: Module 3; Behavioral: Module 4
- Low FODMAP-diet (Active Comparator)
  Interventions: Behavioral: Module 1; Behavioral: Module 2; Behavioral: Module 3; Behavioral: Module 5
- Combined treatment (Active Comparator): Low FODMAP-diet and behavioral therapy
  Interventions: Behavioral: Module 1; Behavioral: Module 2; Behavioral: Module 3; Behavioral: Module 4; Behavioral: Module 5

INTERVENTIONS:
Behavioral: Module 1 — Module 1: Introduction to IBS by a gastroenterologist.
Behavioral: Module 2 — Module 2:Introduction to pain physiology and how the nervous system works by a physiotherapist including practical exercises.
Behavioral: Module 3 — Module 3: Evidence-based guidelines for diet and lifestyle advice (NICE Guidelines) by a clinical dietitian.
Behavioral: Module 4 — Module 4: Intervention: behavioral therapy (exposure therapy and cognitive behavioral therapy).
  Arms: Behavioral therapy; Combined treatment
Behavioral: Module 5 — Module 5: Intervention: The low FODMAP diet.
  Arms: Combined treatment; Low FODMAP-diet

SUMMARY:
The aim of this work is to identify whether the digital treatment program Mage-tarmskolen has an effect on patients with IBS. Our secondary objectives is to address multiple aspects of digital treatmtent success of the different modules. The patients will be randomized to one of four arms and will be delivered different kinds of digital treatment. All patients will have access to ask questions to a registered dietitian. Primary end point is the proportion of patients with treatment success in the low FODMAP, behavioral therapy or both groups, versus the patient education group (sham). Treatment effect is defined as an improvement of 50 points or more on the IBS severity scoring system at 3 months after treatment start compared to the score before treatment.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosed with IBS in the primary or secondary healthcare service.

* Patients aged 18-70 years with IBS defined by the Rome IV criteria: Recurrent abdominal pain, on average at least 1 day per week during the previous 3 months, that is associated with two or more of the following: i) Defecation, either increased pain or pain relief, ii) Change in stool frequency, iii) Change in stool form (appearance)
* All participants >50 years: Colonoscopy within the last 5 years prior to study entry excluding other pathology
* Bank-ID and access to tablet, PC or smart phone.
* No known presence of: symptomatic endometriosis, Diabetes type 1 and 2, Malignant disease (excluding basalioma),
* No history of: severe psychiatric disorder, alcohol or drug abuse, inflammatory bowel disease, microscopic colitis, diverticulitis or ileus, major abdominal surgery (except appendectomy, cholecystectomy, caesarean section, and hysterectomy)
* No "red flags'' indicating severe undiagnosed disease: Night sweats (Repeated episodes of extreme perspiration that may soak nightclothes or bedding), Unintentional weight loss (≥ 4.5 kilograms, or 5% of normal body weight) over less than 6 months without knowing the reason, or blood in stool
* Not pregnant
* Ability to comply with protocol requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 728 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
IBS-SSS | 3 months after treatment start
  Treatment success is defined as an improvement of ≥50 points on the IBS severity scoring system (IBS-SSS) at 3 months after treatment start, compared to the score before treatment

SECONDARY OUTCOMES:
IBS-QOL | 3 months after treatment start
  ≥10-point increase in the IBS-Qualiy of Life (IBS-QoL) at 3 months compared to the score before treatment.
HADS | 3 months after treatment start
  ≥3-point decrease in HADS at 3 months compared to the score before treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Vestlandet, Norway